CLINICAL TRIAL: NCT05830227
Title: Evaluation of Infrared Thermal Imaging in Diagnosis of Obstructive Sleep Apnea Hypopnea Syndrome in Children
Brief Title: Evaluation of Infrared Thermal Imaging in Diagnosis of OSAHS in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Lijun Zeng, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Infrared-thermal-imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary snoring group: Primary snoring group
- Critical OSAHS group: Critical OSAHS group
- Mild OSAHS group: Mild OSAHS group
- Moderate to severe OSAHS group: Moderate to severe OSAHS group

SUMMARY:
OSAHS is a common sleep breathing disorder in children, with the same incidence as childhood asthma, and is mainly caused by upper airway stenosis caused by tonsil/adenoid hyperplasia. Clinical findings show that children with OSAHS often present rhinitis symptoms and like rubbing eyes, but there is no evidence to suggest a correlation. Children with OSAHS suffer from recurrent hypoxemia during sleep, and the existing detection methods such as lateral nasopharyngeal radiographs and electronic nasopharyngoscopy can only reflect the structural and morphological changes of the oral, nasal and pharyngeal tissues, but cannot prove their functional status. Previous studies have found that infrared thermal imaging can reflect the oral, nasal and pharyngeal inflammation of patients, and the infrared expression of patients' frontal region and eyes can also reflect the physiological changes caused by sleep deprivation.

DETAILED DESCRIPTION:
In this project, the children were divided into four groups: primary snoring, critical OSAHS, mild OSAHS and moderate to severe OSAHS, and the tests were completed, including lateral nasopharyngeal radiographs, infrared detection of oropharynx and pharynx, infrared detection of frontal area and eye area, intelligence and behavior scale assessment, etc. Furthermore, the correlation between infrared detection and obstructive sleep apnea hypopnea index, peripheral blood oxygen saturation, adenoid hyperplasia degree of nasopharyngeal lateral film as parameters were analyzed, and the sensitivity and specificity of infrared detection was determined to confirm the diagnostic value of OSAHS. It provides a theoretical basis for finding a convenient, non-damaging, non-radiation, visual and suitable for children functional image detection method.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2 to 14 with SDB related symptoms

Exclusion Criteria:

* 1) Congenital abnormalities of the nose and throat or airway;

  2) craniofacial deformity

  3) Neuromuscular dysregulation

  4) History of adenoids and/or tonsillectomy.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: -Children ages 2 to 14 with SDB related symptoms
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between infrared expression of oral, nasal and pharyngeal inflammation and disease severity | 2025
  Correlation between infrared expression of oral, nasal and pharyngeal inflammation and disease severity (sleep breathing parameters OAHI and LSpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Lijun Zeng [lzeng], Guangdong, Uangdong, China

IPD SHARING:
Plan to Share IPD: No
Observe and study before sharing